CLINICAL TRIAL: NCT00111696
Title: Phase I Study of the Tumor Saturation and Biological Activity of MEDI-522 (Abergrin), a Humanized Monoclonal Antibody Directed Against the Human Alpha V Beta 3 Integrin, in Patients With Advanced Malignant Melanoma
Brief Title: Study of the Tumor Saturation and Biological Activity of MEDI-522 (Abergrin) in Patients With Advanced Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Lawrence Danel-Moore, M.D., PhD, VP, Clin. Dev., MedImmune LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP121; CRRI #0305014 (Other: MedImmune - placeholder); UPCI 05-025 (Other: MedImmune - placeholder)
Record Dates: First submitted 2005-05-24; First posted 2005-05-25 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — etaracizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEDI-522 (Experimental): Drug
  Interventions: Biological: MEDI-522

INTERVENTIONS:
Biological: MEDI-522 — Supplied at a concentration of 50 mg/mL in both 2 mL and 10mL vials

SUMMARY:
To describe the tumor tissue saturation by MEDI-522 in patients with advanced malignant melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable, Stage IV or recurrent malignant melanoma (based on American Joint Committee on Cancer [AJCC] staging)
* Prior therapy with chemotherapy and/or immunotherapy for malignant melanoma is allowed, provided that therapy ended prior to study entry and all treatment related toxicities have resolved
* Measurable disease (based on Response Evaluation Criteria in Solid Tumors [RECIST] criteria) defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques, or as greater than or equal to 10 mm with a spiral computed tomography (CT) scan
* Have melanoma that can be biopsied once before, and at least twice after, MEDI-522 treatment
* Males and females of at least 18 years of age at the time of study entry
* Women of reproductive potential (defined as being <1 year post-menopausal) must have a negative serum B human chorionic gonadotropin (bHCG) pregnancy test within 3 days prior to study entry; and men and women of reproductive potential must agree to practice an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device [IUD], condom, diaphragm with spermicide, cervical cap, abstinence, or sterile sexual partner) at the time informed consent is signed (women only) or at the time of the initiation of MEDI-522 (men only), and must agree to continue using such precautions while receiving MEDI-522 and for 30 days after the final dose of MEDI-522
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 16 weeks
* WBC greater than or equal to 3000/mm(3), absolute neutrophil count (ANC) greater than or equal to 1,500/mm(3), platelet count greater than or equal to 100,000/mm(3)
* Bilirubin greater than or equal to 1.5 mg/dL [unless due to Gilbert's syndrome (unconjugated hyperbilirubinemia) in which case the bilirubin should be <= 3.5 mg/dL]; aspartate transaminase (AST)/alanine transaminase (ALT) greater than or equal to 3 x upper limit of normal (ULN); serum creatinine greater than or equal to 1.5 mg/dL; hepatic alkaline phosphatase greater than or equal to 3.0 x ULN; prothrombin time (PT) or international normalized ratio (INR) within normal range (unless a patient is receiving anticoagulation therapy); or partial thromboplastin time (PTT) within normal range
* Patients who have had prior radiation therapy are eligible, provided that therapy was palliative in nature, not in the area where the tumor will be biopsied, and all radiation-related toxicities have resolved
* Patients who had prior major surgery are eligible if at least 4 weeks have passed since their surgery. All surgical wounds must have healed.
* All toxicities related to prior adjuvant therapy must have resolved.
* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization obtained from the patient prior to receipt of any study medication or beginning study procedures

Exclusion Criteria:

* Pregnancy or nursing
* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for treatment of cancer
* Current or planned participation (from day of study entry through 30 days after last dose of MEDI-522) in a research protocol in which an investigational agent may be administered
* Received an investigational agent within 4 weeks prior to study entry
* Known brain metastases or primary brain tumors
* History of prior malignancies within the past 5 years other than non-melanomatous skin cancers that have been controlled, carcinoma in situ of the cervix, T1a or T1b prostate cancer noted incidentally during a transurethral resection of the prostate (TURP) with prostate-specific antigen (PSA) values within normal limits since TURP, or superficial bladder cancer
* Any evidence of or history, elicited by the investigator, of symptomatic cerebrovascular events (i.e., stroke or transient ischemic attack) within 6 months prior to study entry; or any history or evidence of pulmonary embolism or thrombophlebitis (including deep vein thrombosis) requiring anticoagulant therapy (e.g., warfarin or heparin).
* Currently requiring anticoagulation (excluding use of heparin flush solutions for maintenance of catheter lines) for any thromboembolic disease based on medical history and physical examination
* Any current evidence of hematemesis, melena, hematochezia, or gross hematuria
* History or presence of bleeding diatheses
* Elective surgery planned during the study period through 30 days after the last dose of MEDI-522
* History of hypersensitivity to a previously administered monoclonal antibody
* History of immunodeficiency
* Patients with a clinical diagnosis of Acquired Immune Deficiency Syndrome (AIDS) or known active viral hepatic infections
* A prior myocardial infarction or angina, or uncontrolled/refractory hypertension within 6 months prior to study entry
* Any evidence of an active infection requiring parenteral anti-infective therapy
* Prior treatment with MEDI-522 or MEDI-523
* A general medical or psychological condition or behavior, including substance dependence or abuse that, in the opinion of the investigator, might not permit the patient to complete the study or sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-05; Primary Completion 2007-08 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is to describe the tumor tissue saturation by MEDI-522 in patients with advanced malignant melanoma. | Baseline to disease progression

SECONDARY OUTCOMES:
Describe tumor and endothelial cell viability induced by MEDI-522. | Baseline and two post-therapy points after week 3 and at time of 1st disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Stergios Moschos, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University Of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States